CLINICAL TRIAL: NCT01683539
Title: A Dismantling Study of Cognitive Remediation for Supported Employment
Brief Title: Understanding How Cognitive Remediation Works
Acronym: Cog-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Mcgurk, Associate Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2837E; 2R01MH077210-05A1 (NIH)
Record Dates: First submitted 2012-08-17; First posted 2012-09-12 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Chronic Mental Disorder; Major Depression; Bipolar Disorder
Keywords: Schizophrenia; Chronic Mental Disorder; Employment; Cognitive remediation; Vocational rehabilitation; Brain-derived Neurotrophic Factor (BDNF)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Thinking Skills for Work Program (Experimental): The Thinking Skills for Work Program includes 5 components delivered by a Cognitive Specialist who works collaboratively with the consumer's Employment Specialist: a) assessing the consumer's strengths and weaknesses in cognitive functioning, and analysis of the contribution of cognitive impairments and other factors to job losses and difficulties obtaining a job; b) teaching coping strategies for dealing with cognitive challenges associated with job search or maintaining a job; c) computer cognitive training involving cognitive exercises with a commercially available software program, which is designed to improve the broad range of cognitive skills through a combination of practice and strategy coaching by the Cognitive Specialist; d) job search planning; and e) job support consultation.
  Interventions: Behavioral: The Thinking Skills for Work Program
- The Cognitive Skills for Work Program (Active Comparator): The Cognitive Skills for Work Program includes 4 components delivered by a Cognitive Specialist who works with the consumer's Employment Specialist: a) assessing the consumer's cognitive strengths and weaknesses their relation to job history b) teaching coping strategies for cognitive challenges associated with job search or maintenance c)job search planning, in which the consumer and the Cognitive and Employment Specialists help identify job leads based on the consumer's interests, and identify cognitive coping strategies and supports the consumer may need to succeed at the workplace; and d) job support consultation, in which the Cognitive and Employment Specialists consult with the consumer on additional cognitive coping strategies to enable the consumer to meet the demands of the job.
  Interventions: Behavioral: The Cognitive Skills for Work Program

INTERVENTIONS:
Behavioral: The Thinking Skills for Work Program — The Thinking Skills for Work includes assessment of cognitive strengths and weaknesses and their relationship with work history, computerized cognitive practice, compensatory strategy training, and integration of cognitive and work services.
  Arms: The Thinking Skills for Work Program
Behavioral: The Cognitive Skills for Work Program — The Cognitive Skills for Work includes assessment of cognitive strengths and weaknesses and their relationship with work history, compensatory strategy training, and integration of cognitive and work services.
  Arms: The Cognitive Skills for Work Program

SUMMARY:
This study is aimed at evaluating whether the computer-based cognitive exercises in the Thinking Skills for Work (TSW) program are critical to improving work and cognitive outcomes in consumers with serious mental illness and cognitive impairment enrolled in supported employment (SE), or whether a streamlined version of TSW without this component (the Cognitive Skills for Work (CSW) program) is equally effective for some or all consumers. An RCT will be conducted at two sites (Mental Health Center of Greater Manchester in New Hampshire and Thresholds Inc. in Illinois) with 244 consumers randomly assigned to one of two groups (122 each, with approximately 122 participants having schizophrenia or schizoaffective disorder and 122 of the participants having other diagnoses): 1) TSW, or 2) CSW. The TSW and CSW programs will be delivered by the same Cognitive Specialists, who will work as members of the SE team to integrate cognitive and vocational services. All participants will continue to receive SE services. Participants will be assessed at baseline, post-treatment at 8 months (after completion of the active teaching components of TSW or CSW), and at 16 and 24 months post-baseline to evaluate cognitive functioning, symptoms, and quality of life. All work outcomes will be tracked weekly.

In addition, a supplementary study, commencing in September 2015, will assess a promising biomarker for understanding the mechanisms underlying the effects of cognitive remediation, brain-derived neurotrophic factor (BDNF), in new enrollees in the parent R01 study. This supplement will complement the aims of the parent R01 by shedding light on possible mechanisms related to how TSW works and for whom, thereby informing efforts to refine and improve the program, as well as targeting individuals who fail to benefit. The supplement will take place at the same sites as the parent R01.

DETAILED DESCRIPTION:
Unemployment is a major burden for people with severe mental illness (SMI) such as schizophrenia, with competitive work rates typically between 10-20%. Over the past two decades, supported employment (SE) has been shown to improve competitive work in persons with SMI, and it is now considered an evidence-based practice (EBP). However, there is a need to improve the effectiveness of SE, as 30-60% of consumers work little or not at all, and jobs are often brief and end unsuccessfully. Cognitive remediation, when combined with vocational rehabilitation, has shown promise for improving work outcomes, including in consumers in SE. The most extensively studied approach is the Thinking Skills for Work (TSW) program, developed by this research group, which incorporates computer-based cognitive exercises to restore cognitive skills and teaching compensatory strategies by a Cognitive Specialist who is integrated into the vocational rehabilitation team. Five randomized controlled trials (RCTs), two conducted in SE programs (including one previously conducted by this research group), have shown that adding the TSW program to vocational (SE) services improves work and cognitive outcomes compared to vocational (SE) services alone.

The proposed study takes the next bold step of "dismantling" the TSW program to evaluate whether the cognitive practice exercises component is critical to improving outcomes in SE, or whether a more streamlined and efficient version of the program that focuses only on teaching compensatory skills is sufficient. The study will also yield important information about whether some consumers benefit from computer cognitive exercises, but not others, permitting the TSW program to be individually tailored to consumers' personal needs.

In preparation for the proposed study we developed, standardized, and pilot tested a variant of the TSW program, the Cognitive Skills for Work (CSW) program, that teaches compensatory skills for managing cognitive difficulties but omits computer cognitive exercises, resulting in a program that is approximately one-half the intensity of the original TSW program. A small ongoing pilot study indicated that consumers in SE could be readily engaged and retained in the CSW program and obtain work, supporting the feasibility of this streamlined version of TSW. The proposed research will be an RCT conducted at two high fidelity SE programs, comparing the effects of the TSW and CSW programs in consumers enrolled in SE.

The following hypotheses will be tested:

Primary Hypothesis: Participants in TSW will have better competitive work outcomes than those in the CSW program. This hypothesis is based on the fact that virtually all cognitive remediation research on SMI has included cognitive exercises designed to restore cognitive skills, such as the computer-based cognitive exercises in TSW, with some programs also teaching compensatory strategies. If the null hypothesis is not rejected, and TSW is found to be not significantly more effective than CSW, then dissemination efforts can focus on the more efficient CSW.

Secondary Hypothesis: Participants in TSW will improve more in cognitive functioning than those in CSW. This hypothesis is based on the same rationale as Hypothesis #1.

Exploratory Analyses: In addition to evaluating whether the TSW and CSW programs differ overall in their impact on vocational and cognitive outcomes, we will explore whether consumer characteristics can be identified that predict a differential response to either program. For example, it is possible that consumers with more severe cognitive impairment will respond better to the full TSW program, whereas those with less severe impairment may benefit equally well from the more efficient CSW program.

The proposed research has high potential impact for improving the outcomes of SE, an established EBP for increasing competitive work in SMI, but whose effectiveness is limited by the extent of consumers' cognitive impairment. Maximizing the efficiency of the TSW program, a cognitive remediation program shown to improve work outcomes in two RCTs of SE programs, by determining whether a more streamlined version of the program that requires about one-half the time to implement (the CSW program) is equally effective, could reduce the costs of disseminating and implementing the program, making it accessible to more consumers. This study could also help identify which consumers benefit most from the cognitive exercises component of TSW, thereby facilitating tailoring of the program to the individual's personal needs. Ultimately, this research could play a critical role in making the dream of competitive work a reality for many consumers with SMI.

In addition, a supplementary study, commencing in September 2015, will assess a promising biomarker for understanding the mechanisms underlying the effects of cognitive remediation, brain-derived neurotrophic factor (BDNF), in new enrollees in the parent R01 study. BDNF is a widely distributed protein throughout the central nervous system that promotes neuronal growth and is associated with a broad range of cognitive functions. Limited research suggests that cognitive remediation increases serum BDNF levels, including one study of schizophrenia and another study of Parkinson's disease. This supplemental study will provide a test of whether computerized cognitive training contributes to increased BDNF levels, and whether increases in BDNF are associated with improved cognitive functioning. The supplement will take advantage of the ongoing parent R01 study of the TSW program by measuring BDNF levels at baseline, following delivery of computerized cognitive training/teaching coping skills (6-8 months after baseline), and at two follow-ups (16 and 24 months after baseline) in a diagnostically heterogeneous sample of 38 consumers with impaired cognitive functioning. This supplement will complement the aims of the parent R01 by shedding light on possible mechanisms related to how TSW works and for whom, thereby informing efforts to refine and improve the program, as well as targeting individuals who fail to benefit.

The supplementary study will test the following hypotheses:

Primary Hypothesis: Participants in TSW will show greater increases in BDNF levels from baseline to post-training than participants in CSW. This hypothesis is based on the expectation that the computerized cognitive training exercises in TSW will lead to greater improvements in cognitive functioning than training in compensatory strategies only in CSW, with increases in BDNF levels associated with improved cognitive performance. We also expect that greater increases in BDNF for the TSW group will be maintained at the 16- and 24 month follow-up assessments.

Secondary Hypotheses: 1.) Greater improvements in cognitive functioning from baseline to the post-training and follow-up assessments in TSW than CSW will be associated with stronger increases in BDNF levels over the same assessment points. This hypothesis tests whether greater gains in BDNF levels for TSW mediate the long-term and sustained improvements in cognitive functioning for this program compare to CSW. 2.) Lower baseline BDNF levels will be associated with less gain in cognitive functioning for TSW. This hypothesis tests whether baseline BDNF levels moderate the effectiveness of TSW on improving cognitive functioning, with lower BDNF levels predicting less benefit. BDNF could both be found to be both a mediator and a moderator of the effects of cognitive remediation on improving cognitive functioning.

The supplement will take place at the same sites as the parent R01: Thresholds Inc. in Chicago, and the Mental Health Center of Greater Manchester, NH. Inclusion and exclusion criteria for the supplemental sub-study are identical to those for parent R01 study. As before, pregnancy is not a rule out for participation in the BDNF supplement study. Phlebotomists associated with each site will draw one tablespoon of blood from clients at each assessment timepoint, therefore, a total of up to four (4) tablespoons of blood might be drawn from each client over the course of the study. Drawing BDNF specimens over the full 24-month course of the study will permit researchers to address several important questions regarding the role of BDNF in contributing to neurocognitive functioning, both in response to cognitive remediation as well as how it interacts with cognitive challenging environmental demands-work.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mental disorder
* Minimum age 18.
* Unemployed
* Wants employment
* Must be a recipient of services at one of two participating agencies
* Fluent in English.
* Cognitively impaired, as defined by 1.0 SD below normative scores in memory or executive functioning
* Willing and legally able to provide informed consent to participate in study. Subjects with court appointed legal guardians will be included.

Exclusion Criteria:

-History of neurological conditions that impair cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
AMOUNT OF EMPLOYMENT | 24 MONTHS
  TOTAL HOURS OF EMPLOYMENT FROM BASELINE TO 24 MONTHS. TOTAL WEEKS OF EMPLOYMENT FROM BASELINE TO 24 MONTHS. TOTAL NUMBER OF JOBS HELD FROM BASELINE TO 24 MONTHS.

SECONDARY OUTCOMES:
EXECUTIVE FUNCTIONING AND MEMORY | BASELINE, 8, 16, and 24 months.
  CHANGE FROM BASELINE IN EXECUTIVE FUNCTIONING AND MEMORY AT 8 MONTHS USING THE MATRICS COGNITIVE ASSESSMENT BATTERY.
  CHANGE FROM BASELINE IN EXECUTIVE FUNCTIONING AND MEMORY AT 16 MONTHS USING THE MATRICS COGNITIVE ASSESSMENT BATTERY.
  CHANGE FROM BASELINE IN EXECUTIVE FUNCTIONING AND MEMORY AT 24 MONTHS USING THE MATRICS COGNITIVE ASSESSMENT BATTERY.

OTHER OUTCOMES:
BRAIN-DERIVED NEUROTROPHIC FACTOR (BDNF) - AS PART OF SUPPLEMENTAL SUB-STUDY | BASELINE, 8, 16, and 24 months.
  CHANGE FROM BASELINE IN LEVELS OF BRAIN-DERIVED NEUROTROPHIC FACTOR (BDNF) AT 8 MONTHS USING ABCAM'S BDNF HUMAN ELISA (ENZYME-LINKED IMMUNOSORBENT ASSAY) KIT.
  CHANGE FROM BASELINE IN LEVELS OF BRAIN-DERIVED NEUROTROPHIC FACTOR (BDNF) AT 16 MONTHS USING ABCAM'S BDNF HUMAN ELISA (ENZYME-LINKED IMMUNOSORBENT ASSAY) KIT.
  CHANGE FROM BASELINE IN LEVELS OF BRAIN-DERIVED NEUROTROPHIC FACTOR (BDNF) AT 24 MONTHS USING ABCAM'S BDNF HUMAN ELISA (ENZYME-LINKED IMMUNOSORBENT ASSAY) KIT.

CONTACTS AND LOCATIONS:
Overall Officials: Susan McGurk, Ph.D., Principal Investigator — Center for Psychiatric Rehabilitation, Boston University
Locations (2):
- United States (2):
  - Thresholds, Chicago, Illinois
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire

IPD SHARING:
Plan to Share IPD: No